CLINICAL TRIAL: NCT02929992
Title: Delivery Optimization for Antiretrovial Therapy (The DO ART Study): A Prospective, Interventional, Randomized Study of Community-based ART Initiation, Delivery, and Monitoring in South Africa and Uganda
Brief Title: Delivery Optimization for Antiretroviral Therapy (The DO ART Study)
Acronym: DO ART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Ruanne Barnabas, Assistant Professor, Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 50607
Record Dates: First submitted 2016-07-12; First posted 2016-10-11 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: HIV; ART

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Home ART initiation (Experimental): Participants who are eligible to initiate ART will start in the home and will pick up their medication refills from a mobile van.
  Interventions: Other: ART initiation in the home; Other: Mobile Van Refill and Monitoring
- Hybrid model (Experimental): Participants will be referred to the clinic to initiate ART, once started they will pick up their medication refills from a mobile van.
  Interventions: Other: Mobile Van Refill and Monitoring; Other: Clinic ART Initiation
- Clinic ART initiation, monitoring and resupply (Active Comparator): This is the standard of care arm. Participants will be given a referral to the clinic to initiate ART and will pick up their medication refills from the clinic.
  Interventions: Other: Clinic ART Initiation; Other: Clinic ART Refill and Monitoring

INTERVENTIONS:
Other: ART initiation in the home — Participants initiate ART use in the home without visiting a clinic
  Arms: Home ART initiation
Other: Mobile Van Refill and Monitoring — Participants will pick up their medication refills from the mobile van and have all clinical monitoring conducted in the mobile van.
  Arms: Home ART initiation; Hybrid model
Other: Clinic ART Initiation — Participants are referred to the clinic to initiate ART use
  Arms: Clinic ART initiation, monitoring and resupply; Hybrid model
Other: Clinic ART Refill and Monitoring — Participants will return to the clinic for ART refill and clinical monitoring.
  Arms: Clinic ART initiation, monitoring and resupply

SUMMARY:
The investigators propose the Delivery Optimization for Antiretroviral Therapy Study - The DO ART Study - a prospective randomized study of strategies to optimize community-based ART initiation, monitoring and resupply among HIV-positive persons in South Africa and Uganda. The investigators will work closely with community members, stakeholders, local providers, and the local Department of Health (DoH) to integrate the community-based ART delivery with HIV clinics, pharmacies and labs. Following community sensitization, participants will be recruited through community-based HTC and HIV clinics. HIV-positive persons not engaged in care will receive point-of-care CD4 testing to determine ART eligibility. HIV-positive persons who are eligible for ART by national guidelines will be randomized to one of three ART delivery arms: (i) Home ART initiation and mobile van ART monitoring and resupply, (ii) Hybrid model with clinic ART initiation and mobile van ART monitoring and resupply, and (iii) Clinic ART initiation, monitoring and resupply - the current standard of care (SOC)

DETAILED DESCRIPTION:
Antiretroviral therapy (ART) has tremendous potential to prevent HIV-associated morbidity, mortality and transmission. With reliable ART supply and monitoring, the life expectancy of HIV-positive persons in southern Africa is comparable to that of HIV-negative persons. However, HIV-associated mortality continues to be high among HIV-positive persons not diagnosed and not engaged in care. Of the 35 million persons worldwide who meet WHO (World Health Organization) guidelines for ART, only 15 million are on ART. For already burdened health care systems faced with more than doubling of persons on ART, effective and efficient ART initiation and monitoring strategies are needed. First line ART regimens are once daily oral regimens and well-tolerated, which increases the simplicity of ART delivery in general, including community-based ART delivery a feasible alternative to clinic-based delivery. A priority for optimization of ART delivery is to directly compare and evaluate the impact and cost of community-based ART initiation and resupply to clinic delivery of ART in high prevalence settings in Africa, in order to expand capacity to provide ART coverage.

The investigators have extensive experience with community-based strategies for HIV testing and linkage to care. In a series of studies, the investigators have demonstrated that community-based HIV testing and counseling (HTC) results in >90% knowledge of serostatus and similarly high linkage rates for HIV-positive persons to HIV care. However, the investigators observed bottlenecks within HIV clinics that resulted in delays in ART initiation, particularly for those with higher CD4 counts; only 59% of HIV-positive ART eligible persons were virally suppressed at 12 months, far below the UNAIDS target of 80%. Those findings suggest that community-based strategies for ART initiation and maintenance could address clinic inefficiencies and patient opportunity costs and barriers to optimize ART delivery.

South Africa and Uganda plan to provide decentralized services, including community health workers, CHWs, (known as community health extension workers, CHEWs, in Uganda) conducting HTC and linkage to care and local pharmacy pick-up locations for medication, to meet the challenge of scaling up ART. The investigators proposed Delivery Optimization for Antiretroviral Therapy (The DO ART Study). A rigorous evaluation of an innovative, decentralized ART optimization strategy to safely and cost-effectively deliver ART and monitor viral suppression among HIV-positive persons in South Africa and Uganda. Using a prospective individually-randomized design, the investigators will compare home ART initiation and local mobile van ART resupply to clinic centered care among HIV-positive persons in South Africa and Uganda. Following community sensitization, participants will be recruited through community-based HTC and HIV clinics. HIV-positive persons who are eligible for ART by national guidelines will be randomized to one of three ART delivery arms: (i) Home ART initiation and mobile van ART monitoring and resupply, (ii) A hybrid model of clinic ART initiation with mobile van ART monitoring and resupply, and (iii) Clinic ART initiation, monitoring and resupply - the standard of care (SOC).

The co-primary outcomes are 1) the proportion of HIV-positive persons who initiate ART and achieve viral suppression and 2) cost per HIV-positive person with suppressed HIV viral load at 12 months. The secondary outcomes are safety, social harms, acceptability, the cost-effectiveness of community-based ART delivery, and understanding qualitatively the drivers of engagement in care.

The investigators hypothesize that community-based ART initiation will be acceptable, efficient and improve outcomes, specifically with prompter ART initiation and a higher proportion of HIV-positive persons achieving viral suppression, compared to the standard clinic ART delivery model. Decentralizing HIV care for asymptomatic individuals will expand the overall capacity of the health system to provide care for HIV-positive persons using the existing clinical infrastructure.

ELIGIBILITY:
Inclusion Criteria:

* Reside in the study community for the duration of follow-up
* Able and willing to provide informed consent
* HIV positive and eligible to start ART according to national guidelines
* Not pregnant
* Normal renal function
* Not receiving treatment for active tuberculosis or other opportunistic infections

Exclusion Criteria:

* No separate exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1539 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
HIV viral suppression at 12 months | 12 Months
  Maximize, through community-based ART initiation and maintenance, the proportion of HIV-positive ART eligible persons who achieve viral suppression at 12 months

SECONDARY OUTCOMES:
Measurement of safety across study arms | 1 month, 3 months, 6 months, 9 months, 12 months
  Compare the rates of clinical adverse events across study arms.
Estimate cost-effectiveness of each arm | 12 months
  Estimate the cost-effectiveness for community-based ART initiation compared to clinic-based programs, using mathematical models and study results.
Qualitative review | 1 month, 3 months, 6 months, 9 months, 12 months
  Use qualitative methods to assess "how" and "why" community-based strategies of ART initiation, re-supply and monitoring impact viral suppression and other study outcomes.
Minimize the cost of achieving viral suppression | 12 months
  Minimize the cost per HIV-positive person achieving viral suppression and retention in the continuum of HIV care through community-based strategies compared to clinic standard of care
Measurement of social harms | 12 months
  Compare the rates of reported social harms across study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Ruanne Barnabas, MBChB, DPhil, Principal Investigator — Assistant Professor
Locations (2):
- HSRC Sweetwaters, Sweetwaters, KwaZulu-Natal, South Africa
- ICOBI, Kabwohe, Bushenyi, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barnabas RV, Szpiro AA, van Rooyen H, Asiimwe S, Pillay D, Ware NC, Schaafsma TT, Krows ML, van Heerden A, Joseph P, Shahmanesh M, Wyatt MA, Sausi K, Turyamureeba B, Sithole N, Morrison S, Shapiro AE, Roberts DA, Thomas KK, Koole O, Bershteyn A, Ehrenkranz P, Baeten JM, Celum C; Delivery Optimization of Antiretroviral Therapy (DO ART) Study Team. Community-based antiretroviral therapy versus standard clinic-based services for HIV in South Africa and Uganda (DO ART): a randomised trial. Lancet Glob Health. 2020 Oct;8(10):e1305-e1315. doi: 10.1016/S2214-109X(20)30313-2. PMID 32971053